CLINICAL TRIAL: NCT00797420
Title: Pharmacokinetics of a Fluconazole Loading Dose in Infants and Toddlers
Brief Title: Pharmacokinetics (PK) Study of a Fluconazole Loading Dose in Infants and Toddlers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Benjamin (Other)
Collaborators: Pediatric Pharmacology Research Units Network (Network)
Responsible Party: Sponsor-Investigator, Daniel Benjamin, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011454; NIH-5U10-HD-045962-04
Record Dates: First submitted 2008-11-23; First posted 2008-11-25 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Candidiasis
Keywords: fluconazole; pharmacokinetic; candidiasis; sepsis; pediatric; infants; antifungal; candidemia; fungemia; loading dose
MeSH Terms: conditions — Candidiasis; Sepsis; Candidemia; Fungemia | interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loading Dose (Other): Loading Dose
  Interventions: Drug: Fluconazole Loading Dose
- Loading & high dose (Other): Loading dose & high dose Fluconazole
  Interventions: Drug: Fluconazole Loading Dose & High Dose

INTERVENTIONS:
Drug: Fluconazole Loading Dose — Single Fluconazole loading dose 25 mg/kg
  Other Names: Diflucan
  Arms: Loading Dose
Drug: Fluconazole Loading Dose & High Dose — Fluconazole loading dose 25 mg/kg, followed by fluconazole 12 mg/kg q24 hours for total of 5 days
  Other Names: Diflucan
  Arms: Loading & high dose

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics and safety of a fluconazole loading dose in infants and toddlers.

DETAILED DESCRIPTION:
This is an open label study to investigative the pharmacokinetics and safety of a fluconazole loading dose in infants and toddlers < 2 years of age with suspected sepsis. There will be two treatment groups: single fluconazole loading dose 25 mg/kg; fluconazole loading dose 25mg/kg followed by 12 mg/kg daily for total of 5 days. There will be three age cohorts within each group: pre-term < 30 week EGA infants > 48 hours and < 31 days; > 30 weeks EGA infants > 48 hours and < 31 days; infants ≥ 31 days and < 2 years of age. The study requires administration of fluconazole over 1-5 days depending on treatment group followed by 1 week of safety monitoring. Six to eight 100 µL PK samples will be obtained over the 5 days of drug administration. The risks are reasonable vs. the benefits and have been minimized appropriately. There may be benefit to the subjects (administration of empirical antifungal therapy), and information from the study may benefit a large number of other infants and toddlers with suspected or proven fungal sepsis. There is a data analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* suspected sepsis with blood culture within 48 hours
* age ≥ 48 hours and < 2 years of age
* sufficient venous access to permit study drug administration

Exclusion Criteria:

* allergic reaction to azole
* history of fluconazole administration in prior 5 days
* liver dysfunction
* renal failure
* concomitant use of cyclosporine, tacrolimus, or azithromycin

Ages: 48 Hours to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Fluconazole | 6-8 samples over 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Benjamin, MD, Principal Investigator — Duke University
Locations (1):
- Duke Univeristy Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Benjamin DK Jr, Stoll BJ. Infection in late preterm infants. Clin Perinatol. 2006 Dec;33(4):871-82; abstract x. doi: 10.1016/j.clp.2006.09.005. PMID 17148010
- [Background] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Late-onset sepsis in very low birth weight neonates: the experience of the NICHD Neonatal Research Network. Pediatrics. 2002 Aug;110(2 Pt 1):285-91. doi: 10.1542/peds.110.2.285. PMID 12165580
- [Background] Benjamin DK Jr, DeLong ER, Steinbach WJ, Cotton CM, Walsh TJ, Clark RH. Empirical therapy for neonatal candidemia in very low birth weight infants. Pediatrics. 2003 Sep;112(3 Pt 1):543-7. doi: 10.1542/peds.112.3.543. PMID 12949281
- [Background] Novelli V, Holzel H. Safety and tolerability of fluconazole in children. Antimicrob Agents Chemother. 1999 Aug;43(8):1955-60. doi: 10.1128/AAC.43.8.1955. PMID 10428919
- [Background] Brammer KW, Coates PE. Pharmacokinetics of fluconazole in pediatric patients. Eur J Clin Microbiol Infect Dis. 1994 Apr;13(4):325-9. doi: 10.1007/BF01974613. PMID 8070441
- [Background] Wade KC, Wu D, Kaufman DA, Ward RM, Benjamin DK Jr, Sullivan JE, Ramey N, Jayaraman B, Hoppu K, Adamson PC, Gastonguay MR, Barrett JS; National Institute of Child Health and Development Pediatric Pharmacology Research Unit Network. Population pharmacokinetics of fluconazole in young infants. Antimicrob Agents Chemother. 2008 Nov;52(11):4043-9. doi: 10.1128/AAC.00569-08. Epub 2008 Sep 22. PMID 18809946
- [Background] Anaissie EJ, Kontoyiannis DP, Huls C, Vartivarian SE, Karl C, Prince RA, Bosso J, Bodey GP. Safety, plasma concentrations, and efficacy of high-dose fluconazole in invasive mold infections. J Infect Dis. 1995 Aug;172(2):599-602. doi: 10.1093/infdis/172.2.599. PMID 7622915